CLINICAL TRIAL: NCT04929574
Title: Evaluation of Heart Status in Patients of Beta Thalassemia Using Echocardiogram
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: ZhuHai Hospital (Other); Shenzhen Children's Hospital (Other Government); Shenzhen Second People's Hospital (Other); Jiangmen Maternity and Child Health Care Hospital (Unknown); Yongzhou Maternity and Child Health Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: Heart-Beta thalassemia
Record Dates: First submitted 2021-06-03; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-05

CONDITIONS: Beta Thalassemia
MeSH Terms: conditions — beta-Thalassemia | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- beta thalassemia patients
  Interventions: Diagnostic Test: Echocardiogram and Hematological Analysis

INTERVENTIONS:
Diagnostic Test: Echocardiogram and Hematological Analysis — Echocardiogram and Hematological Analysis

SUMMARY:
Heart failure from myocardial iron deposition is a severe complication for patients with transfusion-dependent beta thalassemia . Increased cardiac iron content impacts the contractility of cardiomyocytes and can also lead to myocarditis, pericarditis, and arrhythmias. The severity of cardiac dysfunction depends on the amount of iron deposited in the myocardium.Echocardiogram is used as noninvasive method to observe heart status. The objective of this study is to evaluate the heart status in patients of Beta Thalassemia from southern China.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with beta-thalassemia

Exclusion Criteria:

* Iron deficiency anemia

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: beta thalassemia patients from Southern China
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Echocardiogram | 3 years
  Evaluation of heart function in beta thalassemia patients by left ventricular fraction shortening

CONTACTS AND LOCATIONS:
Locations (1):
- Southern Medical University, Guangzhou, Guangdong, China